CLINICAL TRIAL: NCT04815109
Title: Prospective Evaluation of Aggravated Sedation in COVID-19 ARDS Patients Using Electroencephalography
Brief Title: Prospective Electroencephalography Evaluation of Sedation in COVID-19
Status: Completed | Type: Observational
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Armin N. Flinspach, Principal Investigator, Goethe University
Other Study IDs: EEG in COVID-19
Record Dates: First submitted 2021-03-23; First posted 2021-03-24 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Conscious Sedation; Pathologic Processes; Electroencephalogram; Acute Respiratory Distress Syndrome; Corona Virus Infection
MeSH Terms: conditions — Pathologic Processes; Respiratory Distress Syndrome; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- critical ill COVID-19: Critically ill COVID-19 patients with need for ventilation and appropriate sedation
  Interventions: Other: Encephalography measurement

INTERVENTIONS:
Other: Encephalography measurement — Encephalography measurement and partially aggravated sedation.

SUMMARY:
Sedation of severe COVID-19 disease are often complicated. We try to find a correlate for this observation by encephalographic studies.

DETAILED DESCRIPTION:
Sedation of critically ill ventilated coronavirus patients, continues to be a challenging issue. Also, neurological symptoms of severe COVID-19 disease have been described frequently. Difficulties in sedation of these patients have been discussed repeatedly. The aim of this study is to investigate whether an encephalographic correlate can be found. Appropriate processed encephalographic techniques have been used for anesthesia monitoring for many years.

The aim of our study is to collect unrelated processed and raw EEG data of sedated COVID-19 patients and to investigate the correlation to the necessary sedation.

ELIGIBILITY:
Inclusion Criteria:

Intubated ventilated patients with SARS-CoV-2 associated acute respiratory distress syndrome and sedation difficulty.

Exclusion Criteria:

Pre-existing severe cerebral brain damage and dysfunction. For example: previous medial infarction, cerebral hemorrhage, structural epilepsy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill COVID-19 patients requiring advanced intensive care treatment with existing intubation-requiring acute respiratory distress syndrome under invasive ventilation. Adequate depth of sedation is usually required for appropriate therapy, which is frequently challenging in COVID-19 patients.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Raw data encephalography measurement | From the beginning of the measurement until the end of the examination (10 to 20 minutes).
  Measurement of the brain activity detectable for the examination procedure in the surface encephalogram.
Processed encephalography measurement | From the beginning of the measurement until the end of the examination (10 to 20 minutes).
  Measurement of detectable algorithm based patient sedation score based on brain activity in the surface encephalogram.

SECONDARY OUTCOMES:
Dosage of continuously administered centrally acting alpha2 agonists. | From 90 minutes before to 10 minutes after encephalographic measurement
  Sedative dosage continuously administered during the measurement interval. [µg/kg/h]
Dosage of continuously delivered central GABA receptor active substances. | From 90 minutes before to 10 minutes after encephalographic measurement
  Sedative dosage continuously administered during the measurement interval. [mg/kg/h]
Dosage of continuously delivered central NMDA receptor active substances. | From 90 minutes before to 10 minutes after encephalographic measurement
  Sedative dosage continuously administered during the measurement interval. [mg/kg/h]
Dosage of continuously delivered opioid based analgesia. | From 90 minutes before to 10 minutes after encephalographic measurement
  Analgetic dosage continuously administered during the measurement interval. [µg/kg/h]

CONTACTS AND LOCATIONS:
Overall Officials: Armin N Flinspach, M.D., Principal Investigator — Goethe-University Frankfurt
Locations (1):
- University Hospital Frankfurt, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analyzed during the current study are not publicly available due to national data protection laws. Upon justified request, the data will be accessible at the primary investigator.